CLINICAL TRIAL: NCT03103958
Title: Phase IV, Double Blind, Randomized, Study Between Probiatop and Placebo for the Assessment of Improving the Gastrointestinal Function and Intestinal Bacterial Flora in Constipated Patients
Brief Title: Effects of Probiotic on Modulation of the Intestinal Microbiota in Constipated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Farmoquimica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FE4-PROBIATOP-PA-14
Record Dates: First submitted 2017-03-17; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Intestinal Bacteria Flora Disturbance; Constipation
Keywords: probiotic; metagenomic; constipation
MeSH Terms: conditions — Constipation | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic (Active Comparator): Probiotic consists of Lactobacillus acidophilus NCFM, Lactobacillus rhamnosus HN001, Lactobacillus paracasei LPC-37 and Bifidobacterium lactis HN019 (Probiatop), Subjects will take two sachets per day after diluting them in 100 ml of water for 28 days.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo consists of maltodextrin. Subjects will take two sachets per day after diluting them in 100 ml of water for 28 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiatop is a live microbial preparation saches containing 1g of the formulation composed by Lactobacillus acidophilus NCFM, 10⁹, Lactobacillus rhamnosus HN001 10⁹, Lactobacillus paracasei LPC-37 10⁹, Bifidobacterium lactis HN019 10⁹ combined with Polydextrose.
  Subjects will take two sachets per day after diluting them in 100 ml of water
  Other Names: Probiatop
  Arms: probiotic
Dietary Supplement: Placebo — The placebo sachets were prepared by substituting equivalent amounts of Maltodextrin for the probiotic powder.
  Subjects will take two sachets per day after diluting them in 100 ml of water
  Arms: Placebo

SUMMARY:
The probiotic for oral use, Probiatop®, consists of Lactobacillus acidophilus NCFM, Lactobacillus rhamnosus HN001, Lactobacillus paracasei LPC-37 and Bifidobacterium lactis HN019. Its activity will be compared with placebo (Maltodextrin). The metagenomics data will be correlated with the Quality of Life Questionnaire answers obtained from participants with intestinal transit problem. The Increase in the number of evacuations, as well as the improvement of complaints related to intestinal transit alteration will be evaluated during the study. The participants will use probiotic or placebo for a period of 28 days and the gastrointestinal function questionnaire and collect stool will be performed before the study and after period of treatment

DETAILED DESCRIPTION:
It is a double-blind, randomized, placebo control study that evaluated the action of a probiotic in relation to a placebo in the human intestinal microbiome by the technique of metagenomics, as well as evaluated the effects of this probiotic on the gastrointestinal transit of constipated participants.

One hundred and twenty constipated patients will be randomized into two groups:Probiatop or Placebo. The first 22 patients from each group will also perform a metagenomic evaluation through the stool sample collection before and after of treatment. Besides these procedures, all patients will fill out a symptom assessment questionnaire at baseline of the study, and then after 14 and 28 days after the beginning of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Agree to adhere to the procedures and requirements of the study and attend the institute on the day (s) and time (s) determined for the evaluations;
* Being able to consent study participation
* Have one or more complaints of change in bowel habits in the last 3 months with onset of symptoms at least 6 months before diagnosis, as described below:

  * Evacuation effort for at least 25% of defecations
  * Lumpy stools, on sausage-shaped or hardened in at least 25% of stools, according to the Bristol scale. number 1, 2 or 3;
  * Incomplete evacuation count in at least 25% of defecations;
  * Feeling of anorectal obstruction / blockage of feces in at least 25% of defecations;
  * Manufactured manuals to facilitate at least 25% of stools (for example, evacuation with digital help, pelvic floor support)

Exclusion Criteria:

* Pregnancy or breast-feeding;
* Known intolerance or allergy to any of the study products;
* Previous history of gastrointestinal surgery;
* Patients with celiac disease or inflammatory bowel disease;
* Patients with psychiatric, cardiologic, respiratory, renal and hepatic disease;
* No acceptance of study admission by the participant; Diagnosis of Clostridium difficile diarrhea in the last 3 months;
* Patients with known immunosuppressive disease;
* Any other gastrointestinal pathology;
* Prior use of antibiotics in less than 30 days;
* Frequent use of laxatives or other medication that alters bowel motility (one week without Use before inclusion)
* Regular treatment with probiotics / symbiotic, including regular use of yogurt with probiotics (One week before use before inclusion)
* Regular use of antidepressant, opioid analgesic, antispasmodic or anticholinergic agents

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2016-08-09 (Actual); Study Completion 2016-09-06 (Actual)

PRIMARY OUTCOMES:
Increased number of bowel movements | 28 days
  Participants will record the number of defecations per day in a daily diary during the study

SECONDARY OUTCOMES:
Incidence of Adverse events | 28 days
  Participants will record the adverse events in a daily diary during study
Changes of intestinal bacteria flora | 28 days
  Quantitative analysis of the participants' microbiota bacteria by sequencing the 16S rDNA gene and the readings obtained from each participant werw compared with genomic banks for identification of the microorganism.
Improve the quality of life of participants evaluated through quality of life questionnaire | 28 days
  The evaluation was performed through quality of life questionnaire.
Evaluation of symptoms of constipation | 28 days
  Improvement of symptoms of constipation by criteria and Bristol scale
Improvement of symptoms of constipation | 28 days
  Improvement of symptoms of constipation by ROME III

CONTACTS AND LOCATIONS:
Overall Officials: Ludmila Donato, Monitor, Study Chair — FQM

IPD SHARING:
Plan to Share IPD: No